CLINICAL TRIAL: NCT01505621
Title: Novel Methodology to Measure Protein Accumulation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Professor of Medicine, Mayo Clinic
Other Study IDs: 11-004969
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Aging
Keywords: Aging; Protein accumulation; Protein damage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — On day one of the study (day of the study drink administration): blood samples and skeletal muscle biopsy (vastus lateralis). Muscle biopsy tissue will be frozen subsequent to collection.
  Week 2 and 3 of the study: blood sample collection Week 4 of the study: blood sample and skeletal muscle (vastus lateralis) biopsy. Muscle biopsy tissue will be frozen subsequent to collection.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Young: Healthy adults 18-30 years old
  Interventions: Other: L[ring-13C6]phenylalanine
- Elderly: Healthy adults greater than 65 years old
  Interventions: Other: L[ring-13C6]phenylalanine

INTERVENTIONS:
Other: L[ring-13C6]phenylalanine — Oral drink composed of essential amino acids including L[ring-13C6]phenylalanine

SUMMARY:
Accumulation of damaged proteins is thought to underlie many degenerative conditions, including aging, diabetes, Alzheimer's disease, cataracts, and others. Over time, proteins can be irreversibly damaged by a variety of factors, such as reactive oxygen species, and without timely degradation they can accumulate and aggregate. We believe this can contribute to the development of chronic degenerative disorders.

The purpose of this study is to develop a novel methodology for measuring protein accumulation and test it in two groups of people: young (18-30 years) and old (≥65 years). This methodology will require that people drink a solution of essential amino acids that includes isotopically labeled L[ring-13C6]phenylalanine. We will then collect blood and muscle samples, to isolate plasma and skeletal muscle proteins. Participants will return to the study center four more times on a weekly interval.

We hypothesize that older proteins, which persisted in circulation and accumulated over time, will have a higher degree of post-translational oxidative damage than newly synthesized proteins.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years
* Age greater than 65 years

Exclusion Criteria:

* Active or uncontrolled cardiovascular disease
* Chronic kidney disease with serum creatinine ≥ 1.4 mg/dL for women and ≥ 1.5 mg/dL for men
* Chronic liver disease (elevation in serum transaminases ≥ 3 times the upper limit of normal)
* Any debilitating chronic illness, including malignancy
* Significant malabsorptive state, including prior gastric bypass surgery or inflammatory bowel disease
* Diabetes mellitus (types 1 or 2) or glucose ≥ 110 mg/dL.
* Obesity (BMI ≥ 31 kg/m2)
* Anticoagulant therapy (warfarin or heparin) or bleeding disorder that increases risk of bleeding during a muscle biopsy.
* Anemia (hemoglobin ≤ 11 g/dL)
* Use of medications known to modulate protein synthesis, mitochondrial function, and/or glucose homeostasis (including β-blockers and corticosteroids).
* Participation in another study where the 13CPhe was administered during the past 6 months.
* Moderate or high level of structured exercise (on average, ≥ 30 minutes per day and ≥ 2 days per week)
* Pregnancy
* Daily use of tobacco products (smoking or chewing); or smoking ≥7 cigarettes per week, on average. Abstinence from tobacco for ≥3 months is required before enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of otherwise healthy participants will be recruited: young (18-30 years) and old (≥65 years). We anticipate screening up to 30 individuals for each group (up to 60 total for study) in order to enroll 12 individuals for each group (24 total for study). A high ratio of screened to enrolled participants is necessary due to exclusion criteria and concern about finding healthy older participants and relatively inactive younger participants. An equal number of participants will be enrolled in each group. We will attempt to have an equal number of men and women.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Isotopic enrichment of plasma and skeletal muscle proteins achieved by oral ingestion of [13C6]-phenylalanine | 3 weeks
  Administration of an oral amino acid mixture containing isotopically-labeled [13C6]-phenylalanine (13C-Phe) will result in 13C-Phe incorporation into newly synthesized proteins. Measuring isotopic enrichment (IE) of 13C-Phe immediately after administration and weekly for 3 consecutive weeks will allow for estimation of protein accumulation.
Degree of post-translational modifications in plasma and muscle proteins | 3 weeks
  The abundance of post-translational modifications of plasma and muscle proteins will be measured using mass spectrometry.

SECONDARY OUTCOMES:
Assess differences in protein accumulation as a function of age | 3 weeks
  Use the newly developed methodology to assess whether otherwise healthy older adults (≥65 years old) have greater accumulation of plasma and muscle proteins compared to healthy young adults (18-30 years old).
Assess differences in protein modification/damage as a function of age | 3 weeks
  The abundance of post-translational modification/damage of plasma and muscle proteins will be measured using mass spectrometry in young (18-30 years old)and older (>65 years old) adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States